CLINICAL TRIAL: NCT07025005
Title: Clinical Study to Evaluate the Possible Role of Fenofibrate in the Prophylaxis From Peripheral Neuropathy Induced by Bortezomib, Lenalidomide and Dexamethasone Protocol in the Treatment of Patients With Multiple Myeloma
Brief Title: Fenofibrate Role in the Prophylaxis From Peripheral Neuropathy Induced by Bortezomib, Lenalidomide and Dexamethasone (VRd) Protocol in the Treatment of Patients With Multiple Myeloma (MM)
Acronym: VRd MM Fibrate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ashraf Mohamed Alaa Mokhtar, Instructor at Clinical Pharmacy Department -Faculty of Pharmacy- Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264MS945/5/25
Record Dates: First submitted 2025-05-31; First posted 2025-06-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Neuropathy; Multiple Myeloma, Neoplasms
Keywords: peripheral neuropathy; multiple myeloma; bortezomib induced peripheral neuropathy (BIPN); Fenofibrate; VRd protocol; lenalidomide
MeSH Terms: conditions — Peripheral Nervous System Diseases; Multiple Myeloma; Neoplasms | interventions — Bortezomib; Lenalidomide; Dexamethasone; Fenofibrate; Tablets

STUDY DESIGN:
Intervention Model Description: At admission, patients will be randomized through sealed envelopes method into two groups to receive either the VRd regimen or the VRd regimen plus fenofibrate 160 mg:
  Group one: (Control group; n=22): which will receive 6 cycles of VRd regimen (each cycle will be given every 28 days).
  Group two: (Fenofibrate group; n=22): which will receive the same regimen plus Fenofibrate 160 mg once daily.
Who Masked: Participant
Masking Description: sealed envelopes method
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fenofibrate group (Active Comparator): 22 participants will receive 6 cycles of (VRd) regimen plus Fenofibrate 160 mg tablet once daily during the period of the 6 cycles.
  Interventions: Drug: Bortezomib + Lenalidomide + Dexamethasone + Fenofibrate 160 mg tablet
- Control group (Other): 22 participants will receive 6 cycles of VRd regimen (each cycle will be given for 28 days)
  Interventions: Drug: Bortezomib + Lenalidomide + Dexamethasone

INTERVENTIONS:
Drug: Bortezomib + Lenalidomide + Dexamethasone + Fenofibrate 160 mg tablet — Bortezomib (VELCADE® 3.5mg/ml) is diluted by 1.4 ml of normal saline (0.9%) solution to give a solution of a concentration of 2.5 mg/mL then the dose will be 1.3 mg/m2 administered subcutaneously at thigh or abdomen at days 1,8,15,22.
  Lenalidomide is given as 25mg orally at days from 1 to 21. Dexamethasone is given as 40mg orally at days 1,8,15,22. Fenofibrate 160 mg tablets orally once daily during the period of the 6 cycles of the(VRd) regimen.
  Arms: Fenofibrate group
Drug: Bortezomib + Lenalidomide + Dexamethasone — Bortezomib (VELCADE® 3.5mg/ml) is diluted by 1.4 ml of normal saline (0.9%) solution to give a solution of a concentration of 2.5 mg/mL then the dose will be 1.3 mg/m2 administered subcutaneously at thigh or abdomen at days 1,8,15,22.
  Lenalidomide is given as 25mg orally at days from 1 to 21. Dexamethasone is given as 40mg orally at days 1,8,15,22.
  Arms: Control group

SUMMARY:
This study aims at evaluating the possible beneficial role of Fenofibrate in attenuating the peripheral neuropathy associated with bortezomib (velcade), lenalidomide (revlimid), and dexamethasone (VRd) regimen in newly diagnosed multiple myeloma patients.The study aims to asses VRd protocol induced peripheral neuropathy through:

1. The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) and The use of Neurotoxicity-12 items questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group "FACT/GOG-Ntx-12 for grading of neuropathy at baseline and by the end of every two VRd cycles.
2. The assessment of biological markers:

Brain -derived neurotrophic factor (BDNF) and Neuro-filament light chain (NfL). through comparing two groups: Group one: (Control group; n=22): which will receive 6 cycles of VRd regimen (each cycle will be given every 28 days).

Group two: (Fenofibrate group; n=22): which will receive the same regimen plus Fenofibrate 160 mg once daily.

DETAILED DESCRIPTION:
Multiple myeloma is considered an incurable disease so several regimens are available for the management of multiple myeloma.

Among these regimens there is the bortezomib, lenalidomide and dexamethasone (RVd or VRd) regimen which is the preferred induction regimen for most patients with newly diagnosed multiple myeloma (NDMM).

Bortezomib has hematologic and non-hematologic adverse reactions. From the non-hematologic adverse reactions there is the bortezomib-induced peripheral neuropathy (BIPN) that remains the most intractable common adverse reactions that occur during bortezomib treatment with no recommended therapies available for preventing or treating existing BIPN.

Fenofibrate a peroxisome proliferator-activated receptor-alpha (PPARα) agonist that is widely used in the management of hypercholesterolemia and hypertriglyceridemia has been proposed as a key lipid metabolism modulator and regulator of inflammation.

Preclinical studies showed that treatment with fenofibrate partially reversed and prevented the development of mechanical and cold hypersensitivity induced by paclitaxel through the regulation of peroxisome proliferator-activated receptor-alpha (PPAR-α) expression and decrease neuroinflammation in the dorsal root ganglia (DRG) without decreasing the antitumoral effect of paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Newly diagnosed MM patients according to the revised International Myeloma Working Group Diagnostic Criteria for the diagnosis of Multiple Myeloma (IMWG).
* Patients being treated by bortezomib-based VRd chemotherapy regimen.
* Patients with performance status <2 according to Eastern Cooperative Oncology Group (ECOG) score.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate liver function (serum bilirubin < 1.2 mg/dl) and adequate renal function (serum creatinine < 1.5 mg/d).

Exclusion Criteria:

* Patients with prior exposure to neurotoxic agents (Cis-platin, vincristine, taxanes, foscarnet, INH, etc..) in the last 6 months.
* Concomitant use of antioxidant vitamins (vitamin A, C, E), anticonvulsants, tricyclic antidepressants, other medications used for neuropathic pain (gabapentin, lamotrigine, carbamazepine).
* Preexisting peripheral neuropathy resulting from other causes such as diabetes and brain disorders, hypothyroidism, autoimmune diseases, hepatitis C.
* Patients with inflammatory diseases (ulcerative colitis, rheumatoid arthritis).
* Patients with conditions associated with oxidative stress (smoking, tuberculosis, comorbid obesity).
* Patients with active liver disease (cirrhosis, fatty liver, hepatitis C, etc..).
* Patients with myopathy.
* Patients with other malignancies.
* Patients with renal impairment, including those with end-stage renal disease and those receiving dialysis.
* Patients with Gallbladder disease and gallstones.
* Pregnant and breast-feeding women.
* Patients with Known allergy to the fenofibrates.
* Concurrent use of statin, colchicine, Ciprofibrate, idelalisib, enzyme inducers (phenytoin, phenobarbitone, carbamazepine,…), enzyme inhibitors (ketoconazole, clarithromycin,…), drugs with high plasma protein binding capacity (Sulfonamides, valproate, oral hypoglycemic, warfarin,…) to avoid potential pharmacodynamics and pharmacokinetic drug interactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in percentage of patients with peripheral neuropathy grade ≥ 2 with the variation of both 12-item neurotoxicity questionnaire (Ntx-12) total score and NCI-CTCAE, v5. | The use of NCI-CTCAE, Version 5, 2017 and "FACT/GOG-Ntx-12" for the grading of peripheral neuropathy will be done at the baseline and by the end of every two VRd cycles ( the duration of each cycle is 28 days) during the 6 VRd cycles duration.
  The change in percentage of patients with peripheral neuropathy grade ≥ 2 using the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5 (NCI-CTCAE, v5) ( where the higher the score the more severity of the peripheral neuropathy) and the use of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity 12 Item Version (FACT/GOG-NTX-12) to assess (where the higher the score, the better the Quality of life).

SECONDARY OUTCOMES:
The change in serum levels of the measured biological markers Brain -derived neurotrophic factor (BDNF) and Neuro-filament light chain (NfL). | The assessment of serum level of the biological markers Brain -derived neurotrophic factor (ng/ml) and Neuro-filament light chain (pg/ml) will be done at the baseline and within 1 week after the 6th VRd cycle ( the duration of each cycle is 28 days).
  The assessment of serum level of the biological markers: Brain -derived neurotrophic factor (BDNF) (in ng/ml) and Neuro-filament light chain (NfL)( in pg/ml) will be done at the baseline (before the initiation of the treatment protocol) and within 1 week after the last VRd cycle (the 6th cycle) ( the duration of each cycle is 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M Alaa, BSc of clinical pharmacy, Principal Investigator — clinical pharmacy departement - Faculty of Pharmacy - Tanta University
Locations (2):
- Egypt (2):
  - Damanhur Oncology Center, Damanhur, El- Behira
  - Tanta University, Tanta, El-Gharbya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin L, Hua H, Ji Y, Jia Z, Peng M, Huang S. Anti-inflammatory role of fenofibrate in treating diseases. Biomol Biomed. 2023 May 1;23(3):376-391. doi: 10.17305/bb.2022.8534. PMID 36724021
- [Background] Azoulay D, Lavie D, Horowitz N, Suriu C, Gatt ME, Akria L, Perlman R, Braester A, Ben-Yehuda D. Bortezomib-induced peripheral neuropathy is related to altered levels of brain-derived neurotrophic factor in the peripheral blood of patients with multiple myeloma. Br J Haematol. 2014 Feb;164(3):454-6. doi: 10.1111/bjh.12624. Epub 2013 Oct 25. No abstract available. PMID 24164472
- [Background] Cebulla N, Schirmer D, Runau E, Flamm L, Gommersbach S, Stengel H, Zhou X, Einsele H, Reinhold AK, Rogalla von Bieberstein B, Zeller D, Rittner H, Kortum KM, Sommer C. Neurofilament light chain levels indicate acute axonal damage under bortezomib treatment. J Neurol. 2023 Jun;270(6):2997-3007. doi: 10.1007/s00415-023-11624-2. Epub 2023 Feb 18. PMID 36802032
- [Background] Caillaud M, Patel NH, White A, Wood M, Contreras KM, Toma W, Alkhlaif Y, Roberts JL, Tran TH, Jackson AB, Poklis J, Gewirtz DA, Damaj MI. Targeting Peroxisome Proliferator-Activated Receptor-alpha (PPAR- alpha) to reduce paclitaxel-induced peripheral neuropathy. Brain Behav Immun. 2021 Mar;93:172-185. doi: 10.1016/j.bbi.2021.01.004. Epub 2021 Jan 9. PMID 33434562
- [Background] Esmaeili MA, Yadav S, Gupta RK, Waggoner GR, Deloach A, Calingasan NY, Beal MF, Kiaei M. Preferential PPAR-alpha activation reduces neuroinflammation, and blocks neurodegeneration in vivo. Hum Mol Genet. 2016 Jan 15;25(2):317-27. doi: 10.1093/hmg/ddv477. Epub 2015 Nov 24. PMID 26604138
- [Background] Yamamoto S, Egashira N. Pathological Mechanisms of Bortezomib-Induced Peripheral Neuropathy. Int J Mol Sci. 2021 Jan 17;22(2):888. doi: 10.3390/ijms22020888. PMID 33477371